CLINICAL TRIAL: NCT00301262
Title: A Multi-Center, Parallel Group, Flexible Dose Trial With A Double-Blind, Randomized, Placebo-Controlled Phase Followed By An Open-Label Phase To Assess The Impact Of Viagra On The Sexual Satisfaction Of Men With Mild Erectile Dysfunction
Brief Title: Impact Of Viagra On Sexual Satisfaction Of Men With Mild Erectile Dysfunction Who Are Sexually Dissatisfied
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481238
Record Dates: First submitted 2006-03-07; First posted 2006-03-10 (Estimated); Results first posted 2008-12-09 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Viagra (Sildenafil citrate)

SUMMARY:
Men's quality of life (QoL) is potentially affected by mild erectile dysfunction (ED) to the same extent as it is by moderate and severe ED. This study will provide controlled clinical data measuring efficacy, QoL parameters and satisfaction changes in men with mild ED treated with Viagra versus those treated with a placebo. With an open-label extension, this study will also provide all study subjects the opportunity to receive the active drug treatment for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men above age of majority
* Mild erectile dysfunction (IIEF-EF 22-25) and sexual dissatisfaction (IIEF-OS 7 or less)

Exclusion Criteria:

* Use of more than 4 doses of any PDE5 inhibitor in the past 12 weeks and use of any PDE5 inhibitor in the past 4 weeks
* Subjects currently taking any other commercially available drug or non-drug treatment for ED

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- Canada (21):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Langley, British Columbia
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Bay Roberts, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, L'Ancienne-Lorette, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Saint-Léonard, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec

REFERENCES:
- [Derived] Kaminetsky JC, Stecher V, Tseng LJ. Quality of erections by age group in men with erectile dysfunction. Int J Clin Pract. 2017 Oct;71(10). doi: 10.1111/ijcp.12976. Epub 2017 Sep 11. PMID 28892218
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481238&StudyName=Impact%20Of%20Viagra%20On%20Sexual%20Satisfaction%20Of%20Men%20With%20Mild%20Erectile%20Dysfunction%20Who%20Are%20Sexually%20Dissatisfied

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 centers in Canada
Pre-assignment Details: 183 subjects entered the study, and 176 subjects were treated in the Double Blind (DB) phase. One subject completed DB phase and continued into the open-label (OL) phase but had no events of sexual activity and therefore, did not take study drug and was excluded from the number of treated subjects, the safety analysis set, and PP population.
Groups:
- DB Viagra / OL Viagra: Subjects started double-blind phase on 50 mg Viagra. After 2 weeks, subjects were allowed to titrate the dose (up or down) depending on efficacy and tolerability and remained on that dose until the end of the double-blind phase (after 8 weeks). Subjects started open-label phase on 50 mg Viagra. After 2 weeks of treatment, subjects were allowed to titrate the dose (up or down) depending on efficacy and tolerability and remained on that dose until the end of open-label phase (after 6 weeks).
- DB Placebo/OL Viagra: Subjects started double-blind phase on matching placebo. After 2 weeks, subjects were allowed to titrate the dose (up or down) depending on efficacy and tolerability and remained on that dose until the end of double-blind phase (after 8 weeks). Subjects started open-label phase on 50 mg Viagra. After 2 weeks of treatment, subjects were allowed to titrate the dose (up or down) depending on efficacy and tolerability and remained on that dose until the end of open-label phase (after 6 weeks).
Period: Double Blind Phase (DB)
Arm/Group | DB Viagra / OL Viagra | DB Placebo/OL Viagra
Started | 94 | 82
Completed | 84 | 69
Not Completed | 10 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Other | 1 | 4
Period: Open Label Phase (OL)
Arm/Group | DB Viagra / OL Viagra | DB Placebo/OL Viagra
Started | 83 | 69
Completed | 79 | 67
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Start : DB Viagra: Subjects started double-blind phase on 50 mg Viagra. After 2 weeks, subjects were allowed to titrate the dose (up or down) depending on efficacy and tolerability and remained on that dose until the end of the double-blind phase (after 8 weeks).
- Start : DB Placebo: Subjects started double-blind phase on matching placebo. After 2 weeks, subjects were allowed to titrate the dose (up or down) depending on efficacy and tolerability and remained on that dose until the end of double-blind phase (after 8 weeks).
- Total: Total of all reporting groups
Arm/Group | Start : DB Viagra | Start : DB Placebo | Total
Number analyzed (Participants) | 94 | 82 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] — DB Viagra/OL Viagra=52.2+/-12.1(n=83) DB Placebo/OL Viagra=48.4+/-12.2(n=69)
  years | 51.6 (12.5) | 48.0 (11.9) | 49.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants] — DB Viagra/OL Viagra Male/Female=83/0 DB Placebo/OL Viagra Male/Female=69/0
  Participants
    Female | 0 | 0 | 0
    Male | 94 | 82 | 176

OUTCOME MEASURES:

1. Primary Outcome: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Index at the End of the DB Treatment (Week 8)
Description: adjusted mean : Possible scores for the EDITS Index range from 0 (extremely low treatment satisfaction) to 100 (extremely high treatment satisfaction).
Time Frame: Week 8
Population: number of subjects in the Full Analysis Set (FAS) population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 88 | 73
scores on a scale | 80.27 (2.329) | 62.15 (2.524)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; The primary analysis population was the FAS. The sample size was estimated based on an expected difference of 16.5 with a standard deviation of 28.4, based on previously observed data; Test type: Superiority or Other; p < 0.0001, ANCOVA — Since there was only one primary endpoint no multiple comparison adjustments were made for primary analysis. Final stat. model included centre, treatment, smoking status and history of ED as factors, and age, duration of ED (baseline) as covariates; Mean Difference (Final Values) = 18.13, 95% CI [11.40 to 24.86], Standard Error of Mean 3.405 — Mean difference between the sidenafil group compared to the placebo group was calculated along with 95% confidence intervals for these differences

2. Secondary Outcome: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Index
Description: Possible scores for the EDITS Index range from 0 (extremely low treatment satisfaction) to 100 (extremely high treatment satisfaction).
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 88 | 80 | 73 | 67
scores on a scale | 79.21 (19.646) | 84.12 (17.220) | 61.64 (22.752) | 87.42 (15.124)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0028, paired t-test; Mean Difference (Net) = 5.09, 95% CI [1.800 to 8.370], Standard Deviation 14.761 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 26.02, 95% CI [20.580 to 31.455], Standard Deviation 22.294 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

3. Secondary Outcome: Change From Baseline to End of Double-Blind Phase (Week 8) in Patient Reported Erectile Function Assessment (PREFA) Total Score
Description: adjusted mean change; PREFA Total Score: 8 = worst; 32 = best.
Time Frame: Week 8
Population: number of subjects in the FAS population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
scores on a scale | 3.97 (0.498) | 2.21 (0.536)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0080, ANCOVA; Mean Difference (Final Values) = 1.76, 95% CI [0.47 to 3.06], Standard Error of Mean 0.656 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Patient Reported Erectile Function Assessment (PREFA) Total Score
Description: PREFA Total Score: 8 = worst, 32 = best.
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra /OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
scores on a scale | 28.54 (3.468) | 29.58 (2.988) | 26.79 (3.753) | 29.73 (2.895)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra /OL Viagra Week 14; Test type: Superiority or Other; p = 0.0051, paired t-test; Mean Difference (Net) = 0.94, 95% CI [0.290 to 1.585], Standard Deviation 2.909 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 2.79, 95% CI [1.812 to 3.770], Standard Deviation 4.013 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

5. Secondary Outcome: Change From Baseline to End of DB Phase (Week 8) in International Index of Erectile Function (IIEF) Domain Scores- Erectile Function
Description: adjusted mean change - Possible total scores for IIEF-EF range from 1 (worst) to 30 (best).
Time Frame: Week 8
Population: number of subjects in the FAS population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
scores on a scale | 2.08 (0.642) | -0.53 (0.698)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0054, ANCOVA; Mean Difference (Final Values) = 2.61, 95% CI [0.78 to 4.43], Standard Error of Mean 0.922 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline to End of DB Phase (Week 8) in International Index of Erectile Function (IIEF) Domain Scores- Orgasmic Function
Description: adjusted mean change - Possible total scores for IIEF-OF range from 0 (worst) to 10 (best).
Time Frame: Week 8
Population: number of subjects in the FAS population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
scores on a scale | 0.59 (0.248) | 0.30 (0.271)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.4232, ANCOVA; Mean Difference (Final Values) = 0.30, 95% CI [-0.43 to 1.02], Standard Error of Mean 0.368 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline to End of DB Phase (Week 8) in International Index of Erectile Function (IIEF) Domain Scores- Sexual Desire
Description: adjusted mean change - Possible total scores for IIEF-SD range from 2 (worst) to 10 (best).
Time Frame: Week 8
Population: number of subjects in the FAS population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
scores on a scale | 0.60 (0.207) | -0.08 (0.223)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0156, ANCOVA; Mean Difference (Final Values) = 0.68, 95% CI [0.13 to 1.22], Standard Error of Mean 0.277 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline to End of DB Phase (Week 8) in International Index of Erectile Function (IIEF) Domain Scores- Intercourse Satisfaction
Description: adjusted mean - Possible total scores for IIEF-IS range from 0 (worst) to 15 (best).
Time Frame: Week 8
Population: number of subjects in the FAS population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
scores on a scale | 2.20 (0.365) | 1.00 (0.390)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0096, ANCOVA; Mean Difference (Final Values) = 1.20, 95% CI [0.30 to 2.11], Standard Error of Mean 0.458 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline to End of DB Phase (Week 8) in International Index of Erectile Function (IIEF) Domain Scores- Overall Satisfaction
Description: adjusted mean change - Possible total scores for IIEF-OS range from 2 (worst) to 10 (best).
Time Frame: Week 8
Population: number of subjects in the FAS population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
scores on a scale | 2.35 (0.254) | 1.46 (0.275)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0135, ANCOVA; Mean Difference (Final Values) = 0.90, 95% CI [0.19 to 1.61], Standard Error of Mean 0.359 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: International Index of Erectile Function (IIEF) Domain Scores- Erectile Function
Description: Possible total scores for IIEF-EF range from 1 (worst) to 30 (best).
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
scores on a scale | 24.92 (5.375) | 26.43 (5.023) | 22.40 (6.403) | 27.67 (3.573)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0033, paired t-test; Mean Difference (Net) = 1.49, 95% CI [0.0510 to 2.465], Standard Deviation 4.392 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 5.22, 95% CI [3.676 to 6.772], Standard Deviation 6.346 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

11. Secondary Outcome: International Index of Erectile Function (IIEF) Domain Scores- Orgasmic Function
Description: Possible total scores for IIEF-OF range from 0 (worst) to 10 (best).
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
scores on a scale | 8.62 (1.812) | 8.95 (1.598) | 7.81 (2.564) | 9.21 (1.213)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.2581, paired t-test; Mean Difference (Net) = 0.20, 95% CI [-0.149 to 0.549], Standard Deviation 1.570 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 1.39, 95% CI [0.758 to 2.018], Standard Deviation 2.582 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

12. Secondary Outcome: International Index of Erectile Function (IIEF) Domain Scores- Sexual Desire
Description: Possible total scores for IIEF-SD and IIEF-OS range from 2 (worst) to 10 (best).
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
scores on a scale | 7.90 (1.665) | 8.10 (1.539) | 7.37 (1.712) | 8.18 (1.230)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.2857, paired t-test; Mean Difference (Net) = 0.18, 95% CI [-0.149 to 0.499], Standard Deviation 1.456 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0005, paired t-test; Mean Difference (Net) = 0.76, 95% CI [0.345 to 1.177], Standard Deviation 1.706 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

13. Secondary Outcome: International Index of Erectile Function (IIEF) Domain Scores- Intercourse Satisfaction
Description: Possible total scores for IIEF-IS range from 0 (worst) to 15 (best).
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
scores on a scale | 11.82 (2.806) | 12.64 (2.367) | 10.84 (2.635) | 13.12 (1.943)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0102, paired t-test; Mean Difference (Net) = 0.75, 95% CI [0.183 to 1.317], Standard Deviation 2.548 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 2.28, 95% CI [1.557 to 3.010], Standard Deviation 2.979 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

14. Secondary Outcome: International Index of Erectile Function (IIEF) Domain Scores- Overall Satisfaction
Description: Possible total scores for IIEF-SD and IIEF-OS range from 2 (worst) to 10 (best).
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
scores on a scale | 8.19 (1.827) | 8.94 (1.656) | 7.25 (2.178) | 9.12 (1.332)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0016, paired t-test; Mean Difference (Net) = 0.68, 95% CI [0.264 to 1.086], Standard Deviation 1.847 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 1.90, 95% CI [1.335 to 2.456], Standard Deviation 2.297 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

15. Secondary Outcome: Change From Baseline to End of DB Phase (Week 8) in Erectile Distress Scale (EDS) Total Score
Description: adjusted mean change - Possible total scores for EDS range from 5 (all of the time) to 30 (none of the time). Higher scores indicate less impact of ED.
Time Frame: Week 8
Population: number of subjects in the FAS population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
scores on a scale | 5.14 (0.870) | 2.36 (0.926)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0083, ANCOVA; Mean Difference (Final Values) = 2.78, 95% CI [0.73 to 4.83], Standard Error of Mean 1.038 — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Erectile Distress Scale (EDS) Total Score
Description: Possible total scores for EDS range from 5 (all of the time) to 30 (none of the time). Higher scores indicate less impact of ED.
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
scores on a scale | 24.58 (6.039) | 24.55 (6.552) | 21.23 (6.246) | 26.58 (4.717)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.9146, paired t-test; Mean Difference (Net) = -0.06, 95% CI [-1.218 to 1.093], Standard Deviation 5.193 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 5.54, 95% CI [3.961 to 7.114], Standard Deviation 6.463 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

17. Secondary Outcome: Change From Baseline to End of DB Phase (Week 8) in Quality of Erection Questionnaire (QEQ) Total Score
Description: adjusted mean change - QEQ raw total score (defined as the sum of scores from QEQ Questions 1 and 3 to 7 and ranged from 6 to 30) was transformed to QEQ total score on a scale of 0 (lowest) to 100 (highest).
Time Frame: Week 8
Population: number of subjects in the FAS population with an observation
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
scores on a scale | 24.04 (3.260) | 5.62 (3.558)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = 18.42, 95% CI [8.88 to 27.96], Standard Error of Mean 4.826 — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Quality of Erection Questionnaire (QEQ) Total Score
Description: QEQ raw total score (defined as the sum of scores from QEQ Questions 1 and 3 to 7 and ranged from 6 to 30) was transformed to QEQ total score on a scale of 0 (lowest) to 100 (highest).
Time Frame: Week 8, Week 14
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
scores on a scale | 80.20 (23.954) | 86.46 (20.918) | 63.64 (28.559) | 89.74 (17.473)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0064, paired t-test; Mean Difference (Net) = 6.41, 95% CI [1.857 to 10.956], Standard Deviation 20.444 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 26.80, 95% CI 2-sided [19.636 to 33.971], Standard Deviation 29.384 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

19. Secondary Outcome: Global Efficacy Question 1 (GEQ1) Response at End of the Double-Blind Phase (Week 8) and at End of the Open-Label Phase (Week 14)
Description: GEQ 1: Compared to having no treatment at all for your erection problem, has the medication you have been taking over the past 4 weeks improved your erections?Responder was defined as answering "Yes". % of responders/non-responders was calculated based on subjects who attempted intercourse.
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Number; unit: percentage of subjects
Arm/Group | Week 8 DB Viagra | Week 8 DB Placebo | Week 14 DB Viagra/OL Viagra | Week 14 DB Placebo/OL Viagra
Number analyzed (Participants) | 88 | 73 | 80 | 67
percentage of subjects
  GEQ1 Responder | 81.8 | 43.8 | 90.0 | 94.0
  GEQ1 Non-Responder | 18.2 | 56.2 | 10.0 | 6.0
Statistical Analysis 1: Comparison: Week 8 DB Viagra vs Week 8 DB Placebo; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 6.491, 95% CI [3.042 to 13.851]

20. Secondary Outcome: Global Efficacy Question 2 (GEQ2) Response at End of the Double-Blind Phase (Week 8) and at End of the Open-Label Phase (Week 14)
Description: GEQ 2: Compared to having no treatment at all for your erection problem, has the medication you have been taking over the past 4 weeks improved your ability to have sexual intercourse? Responder was defined as answering "Yes". % of responders/non-responders was calculated based on subjects who attempted intercourse.
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Number; unit: percentage of subjects
Arm/Group | Week 8 DB Viagra | Week 8 DB Placebo | Week 14 DB Viagra/OL Viagra | Week 14 DB Placebo/OL Viagra
Number analyzed (Participants) | 88 | 73 | 80 | 67
percentage of subjects
  GEQ2 Responder | 79.3 | 45.2 | 86.3 | 92.5
  GEQ2 Non-Responder | 20.7 | 54.8 | 13.8 | 7.5
Statistical Analysis 1: Comparison: Week 8 DB Viagra vs Week 8 DB Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.915, 95% CI [2.396 to 10.080]

21. Secondary Outcome: Global Efficacy Question 3 (GEQ3) Response at End of the Double-Blind Phase (Week 8) and at End of the Open-Label Phase (Week 14)
Description: GEQ 3: When you took a dose of study drug and had sexual stimulation, how often did you get an erection that allowed you to engage in satisfactory sexual intercourse? Resp. was defined as answering almost always or always, most times, or sometimes, and non-resp was defined as answering a few times or almost never or never.
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Number; unit: percentage of subjects
Arm/Group | Week 8 DB Viagra | Week 8 DB Placebo | Week 14 DB Viagra/OL Viagra | Week 14 DB Placebo/OL Viagra
Number analyzed (Participants) | 88 | 73 | 80 | 67
percentage of subjects
  GEQ3 Responders | 94.3 | 81.7 | 95.0 | 98.5
  GEQ3 Non-Responders | 5.7 | 18.3 | 5.0 | 1.5
Statistical Analysis 1: Comparison: Week 8 DB Viagra vs Week 8 DB Placebo; Test type: Superiority or Other; p = 0.0187, Regression, Logistic; Odds Ratio (OR) = 3.676, 95% CI [1.242 to 10.875]

22. Secondary Outcome: Percentage of Occasions of Successful Intercourse (Event Log)
Description: Percentage of occasions at which subjects answered yes to the question, did your erection last long enough to have successful intercourse. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to Week 8
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Groups:
- DB Viagra: Subjects started double-blind phase on 50 mg Viagra. After 2 weeks, subjects were allowed to titrate the dose (up or down) depending on efficacy and tolerability and remained on that dose until the end of the double-blind phase (after 8 weeks)
- DB Placebo: Subjects started double-blind phase on matching placebo. After 2 weeks, subjects were allowed to titrate the dose (up or down) depending on efficacy and tolerability and remained on that dose until the end of double-blind phase (after 8 weeks).
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 88 | 73
percentage of occasions | 73.64 (26.689) | 59.73 (33.332)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0037, independent-samples t-test; Mean Difference (Net) = 13.90, 95% CI [4.59 to 23.22], Standard Error of Mean 4.716 — Independent-samples t-test was used to test mean difference of zero between treatment groups (Viagra - Placebo) at each visit interval

23. Secondary Outcome: Percentage of Occasions of Ejaculation and/or Orgasm (Event Log)
Description: as for outcome 22
Time Frame: Baseline to Week 8
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: Percentage of occasions
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 88 | 73
Percentage of occasions | 74.31 (25.300) | 64.60 (31.903)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0321, independent-samples t-test; Mean Difference (Net) = 9.72, 95% CI [0.84 to 18.60], Standard Error of Mean 4.496 — Mean Difference = Week 8 - Baseline

24. Secondary Outcome: Percentage of Occasions of Successful Intercourse (Event Log)
Description: as for outcome 22
Time Frame: Week 8 to Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra / OL Viagra | DB Placebo/OL Viagra
Number analyzed (Participants) | 80 | 67
percentage of occasions | 79.65 (25.309) | 87.63 (21.936)
Statistical Analysis 1: Comparison: DB Viagra / OL Viagra vs DB Placebo/OL Viagra; Test type: Superiority or Other; p = 0.0427, independent-samples t-test; Mean Difference (Net) = -7.97, 95% CI [-15.68 to -0.27], Standard Error of Mean 3.901 — [estimate comment as in outcome 22, analysis 1]

25. Secondary Outcome: Percentage of Occasions of Ejaculation and/or Orgasm Event Log
Description: as for outcome 22
Time Frame: Week 8 to Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra / OL Viagra | DB Placebo/OL Viagra
Number analyzed (Participants) | 80 | 67
percentage of occasions | 77.69 (25.099) | 85.29 (22.257)
Statistical Analysis 1: Comparison: DB Viagra / OL Viagra vs DB Placebo/OL Viagra; Test type: Superiority or Other; p = 0.0533, independent-samples t-test; Mean Difference (Net) = -7.60, 95% CI [-15.32 to 0.11], Standard Error of Mean 3.903 — [estimate comment as in outcome 22, analysis 1]

26. Secondary Outcome: Change From Baseline to Week 8 in Analog Scales- Firmness
Description: mean change - scale of 0 (worst) to 10 (best).
Time Frame: baseline to Week 8
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
units on a scale | 1.55 (2.023) | 0.38 (1.800)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0002, 2-sample independent t-test; Mean Difference (Net) = 1.1670, 95% CI [0.566 to 1.768], Standard Error of Mean 0.3041 — A 2-sample independent t-test was used to test the difference between treatment for the change between baseline and Week 8 (change = Week 8 - baseline)

27. Secondary Outcome: Change From Baseline to Week 8 in Analog Scales- Maintenance
Description: mean change - scale of 0 (worst) to 10 (best).
Time Frame: baseline to Week 8
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
units on a scale | 1.84 (2.421) | 0.40 (2.152)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0001, 2-sample independent t-test; Mean Difference (Net) = 1.4454, 95% CI [0.727 to 2.164], Standard Error of Mean 0.3638 — [estimate comment as in outcome 26, analysis 1]

28. Secondary Outcome: Change From Baseline to Week 8 in Analog Scales- Reliability
Description: mean change - scale of 0 (worst) to 10 (best).
Time Frame: baseline to Week 8
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
units on a scale | 1.61 (2.795) | 0.42 (2.081)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0032, 2-sample independent t-test; Mean Difference (Net) = 1.1821, 95% CI [0.403 to 1.961], Standard Error of Mean 0.3946 — [estimate comment as in outcome 26, analysis 1]

29. Secondary Outcome: Change From Baseline to Week 8 in Analog Scales- General Sexual Performance
Description: mean change - scale of 0 (worst) to 10 (best)
Time Frame: baseline to week 8
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Viagra | DB Placebo
Number analyzed (Participants) | 89 | 73
units on a scale | 1.72 (2.355) | 0.51 (2.109)
Statistical Analysis 1: Comparison: DB Viagra vs DB Placebo; Test type: Superiority or Other; p = 0.0008, 2-sample independent t-test; Mean Difference (Net) = 1.2123, 95% CI [0.511 to 1.913], Standard Error of Mean 0.3549 — [estimate comment as in outcome 26, analysis 1]

30. Secondary Outcome: Analog Scales- Firmness
Description: mean - scale of 0 (worst) to 10 (best)
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
units on a scale | 7.87 (1.872) | 8.25 (1.932) | 6.60 (2.171) | 8.64 (1.264)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0195, paired t-test; Mean Difference (Net) = 0.39, 95% CI [0.064 to 0.711], Standard Deviation 1.454 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 2.09, 95% CI [1.551 to 2.628], Standard Deviation 2.207 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

31. Secondary Outcome: Analog Scales- Maintenance
Description: mean - scale of 0 (worst) to 10 (best)
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
units on a scale | 7.65 (2.138) | 8.01 (2.155) | 5.99 (2.519) | 8.55 (1.617)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0186, paired t-test; Mean Difference (Net) = 0.40, 95% CI [0.069 to 0.731], Standard Deviation 1.489 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 2.67, 95% CI [2.044 to 3.299], Standard Deviation 2.573 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

32. Secondary Outcome: Analog Scales- Reliability
Description: mean - scale of 0 (worst) to 10 (best)
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
units on a scale | 7.35 (2.360) | 7.96 (2.292) | 6.04 (2.306) | 8.55 (1.550)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0033, paired t-test; Mean Difference (Net) = 0.65, 95% CI [0.223 to 1.077], Standard Deviation 1.917 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 2.61, 95% CI [2.042 to 3.182], Standard Deviation 2.335 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

33. Secondary Outcome: Analog Scales- General Sexual Performance
Description: mean - scale of 0 (worst) to 10 (best)
Time Frame: Week 8, Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Viagra Week 8 | DB Viagra/OL Viagra Week 14 | DB Placebo Week 8 | DB Placebo/OL Viagra Week 14
Number analyzed (Participants) | 89 | 80 | 73 | 67
units on a scale | 7.58 (2.077) | 8.01 (1.978) | 6.53 (2.128) | 8.49 (1.319)
Statistical Analysis 1: Comparison: DB Viagra Week 8 vs DB Viagra/OL Viagra Week 14; Test type: Superiority or Other; p = 0.0143, paired t-test; Mean Difference (Net) = 0.45, 95% CI [0.093 to 0.807], Standard Deviation 1.606 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)
Statistical Analysis 2: Comparison: DB Placebo Week 8 vs DB Placebo/OL Viagra Week 14; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Net) = 1.99, 95% CI [1.454 to 2.516], Standard Deviation 2.178 — A paired t-test was used to examine the within treatment difference between week 8 and week 14 (open label phase)

34. Secondary Outcome: Shift in Responder Rate From Week 8 to Week 14 for Global Efficacy Question (GEQ) 1
Description: GEQ 1: Compared to having no treatment at all for your erection problem, has the medication you have been taking over the past 4 weeks improved your erections? Responder was defined as answering Yes to GEQ 1.
Time Frame: Week 8 to Week 14
Population: number of subjects in the FAS population with an observation: Number of subjects with both Week 8 and Week 14 response to GEQ Question 1 under the treatment.
Measure: Number; unit: subjects
Arm/Group | DB Viagra / OL Viagra | DB Placebo/ OL Viagra
Number analyzed (Participants) | 80 | 67
subjects
  Responder at Week 8 / Responder at Week 14 | 61 | 27
  Responder at Week 8 / Non-Responder at Week 14 | 3 | 0
  Non-Responder at Week 8 / Responder at Week 14 | 11 | 36
  Non-Responder at Week 8 / Non-Responder at Week 14 | 5 | 4
Statistical Analysis 1: Comparison: DB Viagra / OL Viagra; Exact p-values calculated using McNemar's test for difference between Week 8 and Week 14; Test type: Superiority or Other; p = 0.0325, McNemar
Statistical Analysis 2: Comparison: DB Placebo/ OL Viagra; Exact p-values calculated using McNemar's test for difference between Week 8 and Week 14; Test type: Superiority or Other; p < 0.0001, McNemar

35. Secondary Outcome: Shift in Responder Rate From Week 8 to Week 14 for GEQ2
Description: GEQ 2: Compared to having no treatment at all for your erection problem, has the medication you have been taking over the past 4 weeks improved your ability to have sexual intercourse? Responder was defined as answering Yes to GEQ 2.
Time Frame: Week 8 to Week 14
Population: number of subjects in the FAS population with an observation: Number of subjects with both Week 8 and Week 14 response to GEQ Question 2 under the treatment.
Measure: Number; unit: subjects
Arm/Group | DB Viagra / OL Viagra | DB Placebo / OL Viagra
Number analyzed (Participants) | 79 | 67
subjects
  Responder at Week 8 / Responder at Week 14 | 60 | 29
  Responder at Week 8 / Non-Responder at Week 14 | 1 | 0
  Non-Responder at Week 8 / Responder at Week 14 | 8 | 33
  Non-Responder at Week 8 / Non-Responder at Week 14 | 10 | 5
Statistical Analysis 1: Comparison: DB Viagra / OL Viagra; Exact p-values calculated using McNemar's test for difference between Week 8 and Week 14; Test type: Superiority or Other; p = 0.0196, McNemar
Statistical Analysis 2: Comparison: DB Placebo / OL Viagra; Exact p-values calculated using McNemar's test for difference between Week 8 and Week 14; Test type: Superiority or Other; p < 0.0001, McNemar

36. Secondary Outcome: Shift in Responder Rate From Week 8 to Week 14 for GEQ3
Description: GEQ3: When you took a dose of study drug and had sexual stimulation, how often did you get an erection that allowed you to engage in satisfactory sexual intercourse? Responder = almost always or always, most times, or sometimes. Non-responder = a few times (much less than half the time) or almost never or never.
Time Frame: Week 8 to Week 14
Population: number of subjects in the FAS population with an observation: Number of subjects with both Week 8 and Week 14 response to GEQ Question 3 under the treatment.
Measure: Number; unit: subjects
Arm/Group | DB Viagra / OL Viagra | DB Placebo / OL Viagra
Number analyzed (Participants) | 79 | 65
subjects
  Responder at Week 8 / Responder at Week 14 | 74 | 54
  Responder at Week 8 / Non-Responder at Week 14 | 0 | 0
  Non-Responder at Week 8 / Responder at Week 14 | 1 | 10
  Non-Responder at Week 8 / Non-Responder at Week 14 | 4 | 1
Statistical Analysis 1: Comparison: DB Viagra / OL Viagra; Exact p-values calculated using McNemar's test for difference between Week 8 and Week 14; Test type: Superiority or Other; p = 0.3173, McNemar
Statistical Analysis 2: Comparison: DB Placebo / OL Viagra; Exact p-values calculated using McNemar's test for difference between Week 8 and Week 14; Test type: Superiority or Other; p = 0.0016, McNemar

37. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of First Erections Grade 0
Description: Per-patient percentage of hardness of erections:Grade 0 = no erection at all. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline to < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 88 | 74 | 83 | 68
percentage of occasions | 7.09 (13.041) | 12.64 (23.834) | 4.50 (12.217) | 3.12 (9.855)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline to < Week 8; Test type: Superiority or Other; p = 0.0624, Independent-samples t-test; Mean Difference (Net) = -5.55, 95% CI [-11.39 to 0.29], Standard Error of Mean 2.958 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.4523, Independent-samples t-test; Mean Difference (Net) = 1.38, 95% CI [-2.24 to 5.01], Standard Error of Mean 1.835 — [estimate comment as in outcome 22, analysis 1]

38. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of First Erections Grade 1
Description: Per-patient percentage of hardness of erections: Grade 1 = increase in size but not hard. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <= Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 88 | 74 | 83 | 68
percentage of occasions | 3.83 (9.600) | 6.31 (15.144) | 3.48 (14.300) | 1.88 (8.269)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.2081, Independent-samples t-test; Mean Difference (Net) = -2.48, 95% CI [-6.35 to 1.40], Standard Error of Mean 1.962 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.4131, Independent-samples t-test; Mean Difference (Net) = 1.61, 95% CI [-2.26 to 5.48], Standard Error of Mean 1.958 — [estimate comment as in outcome 22, analysis 1]

39. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of First Erections Grade 2
Description: Per-patient percentage of hardness of erections: Grade 2 = hard but not hard enough for penetration. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 88 | 74 | 83 | 68
percentage of occasions | 6.96 (11.858) | 8.72 (15.190) | 4.62 (10.038) | 2.26 (7.813)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.4069, Independent-samples t-test; Mean Difference (Net) = -1.77, 95% CI [-5.97 to 2.43], Standard Error of Mean 2.126 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.1137, Independent-samples t-test; Mean Difference (Net) = 2.37, 95% CI [-0.57 to 5.31], Standard Error of Mean 1.489 — [estimate comment as in outcome 22, analysis 1]

40. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of First Erections Grade 3
Description: Per-patient percentage of hardness of erections: Grade 3 = hard enough for penetration but not completely hard. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 88 | 74 | 83 | 68
percentage of occasions | 34.94 (29.253) | 47.17 (32.167) | 29.50 (28.515) | 30.12 (31.412)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.0123, Independent-samples t-test; Mean Difference (Net) = -12.23, 95% CI [-21.77 to -2.70], Standard Error of Mean 4.829 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.8993, Independent-samples t-test; Mean Difference (Net) = -0.62, 95% CI [-10.27 to 9.03], Standard Error of Mean 4.883 — [estimate comment as in outcome 22, analysis 1]

41. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of First Erections Grade 4
Description: Per-patient percentage of hardness of erections: Grade 4 = completely hard. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 88 | 74 | 83 | 68
percentage of occasions | 47.19 (35.293) | 25.16 (33.764) | 57.89 (35.934) | 62.63 (35.112)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p < 0.0001, Independent-samples t-test; Mean Difference (Net) = 22.03, 95% CI [11.25 to 32.81], Standard Error of Mean 5.458 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.4165, Independent-samples t-test; Mean Difference (Net) = -4.74, 95% CI [-16.24 to 6.76], Standard Error of Mean 5.818 — [estimate comment as in outcome 22, analysis 1]

42. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of First Erections Grade 3 or 4
Description: Per-patient percentage of hardness of erections: Grade 3 = hard enough for penetration but not completely hard, Grade 4 = completely hard. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 88 | 74 | 83 | 68
percentage of occasions | 82.13 (23.476) | 72.33 (31.798) | 87.39 (22.496) | 92.75 (15.386)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.0257, Independent-samples t-test; Mean Difference (Net) = 9.80, 95% CI [1.21 to 18.39], Standard Error of Mean 4.351 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.0971, Independent-samples t-test; Mean Difference (Net) = -5.36, 95% CI [-11.70 to 0.98], Standard Error of Mean 3.209 — [estimate comment as in outcome 22, analysis 1]

43. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of Second Erections Grade 0
Description: Per-patient percentage of hardness of second erections: Grade 0 = no erection at all. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 73 | 38 | 61 | 51
percentage of occasions | 0.00 (0.000) | 3.18 (15.052) | 0.13 (0.985) | 2.17 (14.014)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.0726, Independent-samples t-test; Mean Difference (Net) = -3.18, 95% CI [-6.66 to 0.30], Standard Error of Mean 1.754 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.2581, Independent-samples t-test; Mean Difference (Net) = -2.04, 95% CI [-5.61 to 1.52], Standard Error of Mean 1.798 — [estimate comment as in outcome 22, analysis 1]

44. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of Second Erections Grade 1
Description: Per-patient percentage of hardness of second erections: Grade 1 = increase in size but not hard. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 73 | 38 | 61 | 51
percentage of occasions | 6.43 (22.211) | 7.47 (22.317) | 1.70 (9.143) | 2.03 (8.638)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.8158, Independent-samples t-test; Mean Difference (Net) = -1.04, 95% CI [-9.86 to 7.78], Standard Error of Mean 4.450 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.8464, Independent-samples t-test; Mean Difference (Net) = -0.33, 95% CI [-3.68 to 3.02], Standard Error of Mean 1.692 — [estimate comment as in outcome 22, analysis 1]

45. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of Second Erections Grade 2
Description: Per-patient percentage of hardness of second erections:Grade 2 = hard but not hard enough for penetration. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 73 | 38 | 61 | 51
percentage of occasions | 14.93 (28.145) | 15.27 (30.431) | 11.96 (24.555) | 12.66 (28.294)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.9529, Independent-samples t-test; Mean Difference (Net) = -0.34, 95% CI [-11.82 to 11.13], Standard Error of Mean 5.789 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.8899, Independent-samples t-test; Mean Difference (Net) = -0.69, 95% CI [-10.59 to 9.20], Standard Error of Mean 4.994 — [estimate comment as in outcome 22, analysis 1]

46. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of Second Erections Grade 3
Description: Per-patient percentage of hardness of second erections:Grade 3 = hard enough for penetration but not completely hard. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 73 | 38 | 61 | 51
percentage of occasions | 37.41 (38.658) | 47.59 (41.025) | 42.97 (38.322) | 33.29 (31.633)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.2001, Independent-samples t-test; Mean Difference (Net) = -10.18, 95% CI [-25.83 to 5.47], Standard Error of Mean 7.897 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.1527, Independent-samples t-test; Mean Difference (Net) = 9.68, 95% CI [-3.64 to 23.01], Standard Error of Mean 6.724 — [estimate comment as in outcome 22, analysis 1]

47. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of Second Erections Grade 4
Description: Per-patient percentage of hardness of second erections:Grade 4 = completely hard. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 73 | 38 | 61 | 51
percentage of occasions | 41.23 (41.013) | 26.49 (34.300) | 43.24 (39.891) | 49.86 (36.921)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.0606, Independent-samples t-test; Mean Difference (Net) = 14.74, 95% CI [-0.67 to 30.15], Standard Error of Mean 7.774 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.3678, Independent-samples t-test; Mean Difference (Net) = -6.62, 95% CI [-21.12 to 7.88], Standard Error of Mean 7.318 — [estimate comment as in outcome 22, analysis 1]

48. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Hardness of Second Erections Grade 3 or 4
Description: Per-patient percentage of hardness of second erections: Grade 3 = hard enough for penetration but not completely hard, Grade 4 = completely hard. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 73 | 38 | 61 | 51
percentage of occasions | 78.64 (35.395) | 74.08 (40.922) | 86.21 (27.647) | 83.14 (31.561)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.5429, Independent-samples t-test; Mean Difference (Net) = 4.56, 95% CI [-10.25 to 19.37], Standard Error of Mean 7.474 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.5849, Independent-samples t-test; Mean Difference (Net) = 3.07, 95% CI [-8.02 to 14.15], Standard Error of Mean 5.595 — [estimate comment as in outcome 22, analysis 1]

49. Secondary Outcome: Baseline to <Week 8 and Week 8 to <=Week 14 in Event Log: Frequency of Second Erections
Description: Percentage of occasions at which second erection was achieved. Calculation for each subject for each event log endpoint: percentage = (number of occasions with an answer of 'Yes' within visit interval) / (number of occasions within visit interval) x 100.
Time Frame: Baseline to <Week 8 and Week 8 to <=Week 14
Population: number of subjects in the FAS population with an observation
Measure: Mean (Standard Deviation); unit: percentage of occasions
Arm/Group | DB Viagra Baseline < Week 8 | DB Placebo Baseline < Week 8 | DB Viagra/OL Viagra Week 8 to <=Week 14 | DB Placebo/OL Viagra Week 8 to <=Week 14
Number analyzed (Participants) | 88 | 74 | 83 | 68
percentage of occasions | 38.06 (33.287) | 19.20 (28.977) | 44.07 (38.632) | 39.15 (37.159)
Statistical Analysis 1: Comparison: DB Viagra Baseline < Week 8 vs DB Placebo Baseline < Week 8; Test type: Superiority or Other; p = 0.0002, Independent-samples t-test; Mean Difference (Net) = 18.86, 95% CI [9.08 to 28.64], Standard Error of Mean 4.952 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: DB Viagra/OL Viagra Week 8 to <=Week 14 vs DB Placebo/OL Viagra Week 8 to <=Week 14; Test type: Superiority or Other; p = 0.4290, Independent-samples t-test; Mean Difference (Net) = 4.93, 95% CI [-7.35 to 17.20], Standard Error of Mean 6.212 — [estimate comment as in outcome 22, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.